CLINICAL TRIAL: NCT04594759
Title: Weekly Isotretinoin Therapy for the Treatment of Moderate Acne Vulgaris
Brief Title: Weekly Isotretinoin Therapy Study
Acronym: WIT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Samantha Karlin, MD, Dermatology Resident Principal Investigator, Medical University of South Carolina
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00103493
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin

STUDY DESIGN:
Masking Description: The study member assessing change in acne using the Comprehensive Acne Severity Scale does not know the medication the participants are taking.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Drug: Isotretinoin

INTERVENTIONS:
Drug: Isotretinoin — Participants will be getting isotretinoin (1-1.5 mg/kg/week)

SUMMARY:
In current Dermatology practice, options for moderate acne vulgaris remain limited. The mainstay of treatment for moderate acne remains long courses of oral antibiotics despite emerging antibiotic resistance. The efficacy of daily to twice daily dosed isotretinoin, an oral vitamin A derivative, for treatment of severe acne has been well established. The purpose of this study is to determine if once weekly dosed isotretinoin is effective for the treatment of patients with moderate acne. Additionally, the study aims to evaluate patient satisfaction and identify any adverse effects on this alternative dosing regimen.

DETAILED DESCRIPTION:
In current Dermatology practice, options for moderate acne vulgaris remain limited. Moderate acne is clinically defined as acne that has not responded to at least three months of topical therapy and is not severe enough for initial treatment with a conventional course of isotretinoin (formerly known as Accutane). The mainstay of treatment for moderate acne remains long courses of oral antibiotics, mainly tetracyclines (doxycycline, minocycline) and occasionally trimethoprim-sulfamethoxazole. Males with moderate acne, in particular, are especially limited in their treatment options as they are not eligible for hormonal management (spironolactone, oral contraceptive pills) like their female counterparts. Additionally, even for those regardless of gender who may eventually qualify for a traditional isotretinoin course, many insurance companies first require failure to respond to at least three months of oral antibiotics. Nagler et. al found that the average antibiotic use for moderate to severe acne prior to receiving isotretinoin was 331 days, with 15.3% of patients prescribed antibiotics for three months or less, 88% for six months or more, and 46% for at least one year.1 Despite the widespread use of oral antibiotics in acne, antibiotic resistance is considered a global threat per the CDC2, and there have been calls to limit their use in acne because of concerns of bacterial resistance3,4,5. Because of this, there is a significant need for more research on alternative treatment options for moderate acne.

Once weekly isotretinoin dosing has the potential to significantly improve moderate acne with good patient satisfaction and safety profile; however, no study findings on this treatment option have been published to date. The efficacy of isotretinoin, an oral vitamin A derivative, for treatment of acne has been well established. The traditional treatment course for severe acne consists of once to twice daily dosing (0.5-1 mg/kg/day) for 4-7 months (or 150mg/kg total cumulative dose). Though efficacious, there are numerous reported side-effects due to achieving the cumulative dose rapidly by once to twice daily dosing, such as severe dry skin, lips, and eyes, as well as liver enzyme and lipid abnormalities. Because of this, there have been studies exploring alternative isotretinoin dosing regimens including microdose, lower daily dose regimens (0.15-0.4 mg/kg/day6, 0.25-0.4 mg/kg/day7, 0.3-0.4 mg/kg/day8,9, in addition to 5 mg/day10 and 0.15-0.28 mg/kg/day with additional of local application of 1% clindamycin gel every other day11) and daily dosing for 7-10 consecutive days (0.5-0.7 mg/kg/day) out of each month only.7,12,13,14 All studies had favorable outcomes with alternative dosing, despite the lower total cumulative dose versus conventional dosing. Those who also analyzed adverse effect rates with alternative isotretinoin dosing found that these were either rarely observed or similar to conventional dosing.6,8,9,10,12,14 In contrast, the potential adverse effects of oral antibiotics used for acne include photosensitivity and nausea/vomiting (doxycycline), drug-induced pigment deposition and drug-induced systemic lupus erythematosus (minocycline), and angioedema and drug rashes including drug reaction with eosinophilia and systemic symptoms (DRESS) syndrome (trimethoprim-sulfamethoxazole). Interestingly, rates of acne recurrence between alternative isotretinoin dosing and conventional dosing were similar at follow-up,6,7,9 despite a much older study from 1984 that found otherwise.15 Additionally, cost of alternative isotretinoin dosing was lower than with conventional dosing,8,9,13 and patient satisfaction was highest in the alternative dosing groups.7,10 For these reasons, this study aims to evaluate the efficacy of once weekly isotretinoin dosing (1-1.5 mg/kg/week) as a potential alternative to oral antibiotics for the treatment of patients with moderate acne. Secondary endpoints include patient satisfaction and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* All patients 12 years and older with the diagnosis of moderate acne vulgaris

Exclusion Criteria:

* Patients who are at baseline on long-term tetracycline antibiotics, long-term trimethoprim-sulfamethoxazole, or on spironolactone for any reason
* Patients who have taken isotretinoin in the past 6 months
* Patients with hypersensitivity to isotretinoin or to any of its components
* Females who are pregnant, likely to become pregnant, or will be breast-feeding during the study period
* Patients with a history of major depression, mania, or psychosis with an active episode during the past year including current psychotic symptoms and/or current suicidal ideation
* Adult patients with cognitive impairment
* Patients with baseline kidney or liver disease
* Patients with baseline hypertriglyceridemia
* Patients with history of or current pseudotumor cerebri
* Patients with any clinically significant unstable medical condition which could pose a risk to the safety of the patient
* Inability or unwillingness of subject or legal guardian/representative to give informed consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Karlin, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Samantha Karline, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data collected during the study after de-identification
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Immediately following publication, indefinitely

REFERENCES:
- [Background] Nagler AR, Milam EC, Orlow SJ. The use of oral antibiotics before isotretinoin therapy in patients with acne. J Am Acad Dermatol. 2016 Feb;74(2):273-9. doi: 10.1016/j.jaad.2015.09.046. Epub 2015 Oct 30. PMID 26525749
- [Background] Center for Disease Control (https://www.cdc.gov/drugresistance/biggest-threats.html?CDC_AA_refVal=https%3A%2F%2Fwww.cdc.gov%2Fdrugresistance%2Fbiggest_threats.html)
- [Background] Dreno B, Thiboutot D, Gollnick H, Bettoli V, Kang S, Leyden JJ, Shalita A, Torres V; Global Alliance to Improve Outcomes in Acne. Antibiotic stewardship in dermatology: limiting antibiotic use in acne. Eur J Dermatol. 2014 May-Jun;24(3):330-4. doi: 10.1684/ejd.2014.2309. PMID 24721547
- [Background] Bowe WP. Antibiotic resistance and acne: where we stand and what the future holds. J Drugs Dermatol. 2014 Jun;13(6):s66-70. PMID 24918574
- [Background] Ross JI, Snelling AM, Carnegie E, Coates P, Cunliffe WJ, Bettoli V, Tosti G, Katsambas A, Galvan Perez Del Pulgar JI, Rollman O, Torok L, Eady EA, Cove JH. Antibiotic-resistant acne: lessons from Europe. Br J Dermatol. 2003 Mar;148(3):467-78. doi: 10.1046/j.1365-2133.2003.05067.x. PMID 12653738
- [Background] Mandekou-Lefaki I, Delli F, Teknetzis A, Euthimiadou R, Karakatsanis G. Low-dose schema of isotretinoin in acne vulgaris. Int J Clin Pharmacol Res. 2003;23(2-3):41-6. PMID 15018017
- [Background] Lee JW, Yoo KH, Park KY, Han TY, Li K, Seo SJ, Hong CK. Effectiveness of conventional, low-dose and intermittent oral isotretinoin in the treatment of acne: a randomized, controlled comparative study. Br J Dermatol. 2011 Jun;164(6):1369-75. doi: 10.1111/j.1365-2133.2010.10152.x. Epub 2011 May 17. PMID 21114478
- [Background] Amichai B, Shemer A, Grunwald MH. Low-dose isotretinoin in the treatment of acne vulgaris. J Am Acad Dermatol. 2006 Apr;54(4):644-6. doi: 10.1016/j.jaad.2005.11.1061. PMID 16546586
- [Background] Kotori MG. Low-dose Vitamin "A" Tablets-treatment of Acne Vulgaris. Med Arch. 2015 Feb;69(1):28-30. doi: 10.5455/medarh.2015.69.28-30. Epub 2015 Feb 21. PMID 25870473
- [Background] Rademaker M, Wishart JM, Birchall NM. Isotretinoin 5 mg daily for low-grade adult acne vulgaris--a placebo-controlled, randomized double-blind study. J Eur Acad Dermatol Venereol. 2014 Jun;28(6):747-54. doi: 10.1111/jdv.12170. Epub 2013 Apr 26. PMID 23617693
- [Background] Sardana K, Garg VK, Sehgal VN, Mahajan S, Bhushan P. Efficacy of fixed low-dose isotretinoin (20 mg, alternate days) with topical clindamycin gel in moderately severe acne vulgaris. J Eur Acad Dermatol Venereol. 2009 May;23(5):556-60. doi: 10.1111/j.1468-3083.2008.03022.x. Epub 2009 Jan 9. PMID 19143903
- [Background] Akman A, Durusoy C, Senturk M, Koc CK, Soyturk D, Alpsoy E. Treatment of acne with intermittent and conventional isotretinoin: a randomized, controlled multicenter study. Arch Dermatol Res. 2007 Dec;299(10):467-73. doi: 10.1007/s00403-007-0777-2. Epub 2007 Aug 21. PMID 17710426
- [Background] Goulden V, Clark SM, McGeown C, Cunliffe WJ. Treatment of acne with intermittent isotretinoin. Br J Dermatol. 1997 Jul;137(1):106-8. PMID 9274635
- [Background] Kaymak Y, Ilter N. The effectiveness of intermittent isotretinoin treatment in mild or moderate acne. J Eur Acad Dermatol Venereol. 2006 Nov;20(10):1256-60. doi: 10.1111/j.1468-3083.2006.01784.x. PMID 17062042
- [Background] Strauss JS, Rapini RP, Shalita AR, Konecky E, Pochi PE, Comite H, Exner JH. Isotretinoin therapy for acne: results of a multicenter dose-response study. J Am Acad Dermatol. 1984 Mar;10(3):490-6. doi: 10.1016/s0190-9622(84)80100-0. PMID 6233335

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group
Started | 22
Completed | 19
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.77 (8.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Showed Improvement in Their Visible Acne (Efficacy of Once Weekly Isotretinoin)
Description: Will look at clinical photos before, during, and after treatment and grade acne using a validated, clinical grading system (Comprehensive Acne Severity Scale, CASS) with "0" being clear skin and "5" being very severe acne. Participants are eligible for the study if their score is 3 or higher. An improvement in their visible acne is a score of 2, 1, or 0 at the end of the 4 months of treatment.
Time Frame: Baseline and end of treatment, approximately 4 months
Population: The amount of participants that were analyzed is less than the original number enrolled. There were 3 participants that did not complete the study and were not analyzed at the end of the 4 months of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
Participants | 18

2. Secondary Outcome: Number of Participants With a Change in Quality of Life
Description: Participants will use the Dermatology Life Quality Index survey which measures how much their skin problems affect their life. 10 questions are asked with answers "Very much," " A lot," "A little," "Not at all," or "Not relevant". The answers correlate to a number ("Very much" =3, " A lot" = 2, "A little"=1, "Not at all"= 0, "Not relevant"=0) and the answered are added together to get a score for that month. The higher the score the more their skin impacts their day to day activities. An improvement in their quality of life is a lower score at 4 months compared to baseline score.
Time Frame: Baseline, monthly, and end of treatment, total of 4 months
Population: Three subjects did not complete the study for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
Participants | 17

3. Secondary Outcome: Number of Side Effects Reported at the End of 4 Months
Description: Participants will fill out a survey regarding nonserious and serious adverse events.
Time Frame: through study completion, an average of 4 months
Population: 3 participants were lost to follow up and did not complete the final adverse event questionnaire. One participant can have more than one event.
Measure: Number; unit: events
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
events | 24

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 4 months. Participants could have more than one adverse event.
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 12/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=19)
Dry lips/eyes (Skin and subcutaneous tissue disorders) | 10
Dry skin (Skin and subcutaneous tissue disorders) | 11
Mild myalgias (Musculoskeletal and connective tissue disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT04594759/Prot_001.pdf